CLINICAL TRIAL: NCT05090397
Title: Applied Strategies for MRI-Guided High-Definition tDCS for Major Depression
Brief Title: MRI-Guided High-Definition Transcranial Direct Current Stimulation (tDCS) for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amber Leaver, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00213826
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) uses a mild electrical current to make small (or subtle) changes to how the brain works (or functions).
  Arms: Active
Device: Sham Transcranial Direct Current Stimulation — Sham Transcranial Direct Current Stimulation
  Arms: Sham

SUMMARY:
The purpose of this research is to understand how a neurostimulation technique, transcranial electrical stimulation (tES), affects brain function in adults with major depression measured with functional magnetic resonance imaging (fMRI). This study targets a specific kind of tES called transcranial direct current stimulation (tDCS), where a mild, constant current is passed between electrodes placed on the scalp.

DETAILED DESCRIPTION:
This is an investigator-initiated MRI research study of a noninvasive neurostimulation technique, transcranial direct current stimulation (tDCS) using focal "high definition" (HD) electrodes positioned using pre-treatment MRI. Primary objective is to measure changes in brain function during MRI-guided HDtDCS with MRI. Secondary objective is to measure changes in depressive symptoms after five consecutive days of MRI-guided tDCS (20 minutes per session).

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages between 18 and 65
* 2. Race/ethnicity: all races and ethnic groups
* 3. Sex/Gender: all
* 4. Capacity to provide informed consent
* 5. Diagnosis of Major Depressive Disorder made by volunteer's physician at least one year prior (confirmed by patient self-report)
* 6. Currently under the care of a clinician for depression (psychiatrist, psychologist, or other clinician)
* 7. Currently experiencing symptoms of depression (Patient Health Questionnaire 9, PHQ9 >4 at screening; Hamilton Depression Rating Scale 17-item, HDRS-17, score >8 at Visit 1)
* 8. Stable or no pharmacological antidepressant regimen (SSRI, SNRI, MOAI, or tricyclic/TCA) with no change in treatment 6 weeks prior to study start

Exclusion Criteria:

* 1. Ages below 18 (neurobiology is quite different in children vs. adults)
* 2. Ages above 65 (cortical excitability changes with age)
* 3. Active suicidal thoughts, ideation, or behavior with plan within the past month (HDRS-17 item 3 score 3-4)
* 4. Change in antidepressant medication within 6 weeks of study start
* 5. Diagnosis of any medical condition potentially affecting brain function: neuropsychiatric or mental disorders, other mood disorders (bipolar disorder, primary anxiety disorder, PTSD), psychotic states or disorders, developmental disorders, neurological disorders, including mild cognitive impairment, significant head injury, significant history of alcohol/substance abuse or dependence within past 12 months, chronic pain (current, or for more than one year within the past one year), other major medical conditions (e.g., cancer, stroke).
* 6. MRI contraindications: metal or other implants that are not MR-safe, claustrophobia, pregnancy or suspected pregnancy
* 7. tES contraindications: skin conditions or injuries on the scalp hair extensions, wigs, braids, etc. that cannot be removed prior to the study, metal implants or pacemakers (also contraindicated for MRI)
* 8. Non-English speakers (due to written consent and questionnaires administered)
* 9. Neurostimulation or neuromodulation treatment for any reason within the past 3 months
* 10. Current medication use potentially affecting brain function, including decongestants, antihistamines, benzodiazepines or other anticonvulsants, anti-psychotics.
* 11. Prisoners will not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in brain functional connectivity | Acute/immediate
  Functional MRI will measure changes in brain function during tDCS. Specifically, the investigators will measure change in functional connectivity of prefrontal cortex (% change in Fisher's z).

SECONDARY OUTCOMES:
Changes in depressive symptoms (Hamilton) | 1 week, 2 weeks, 1 month
  Symptoms of depression will be measured before and after 5 sessions of tDCS using Hamilton Depression Rating Scale (HDRS 17-item). Change HDRS score will be used as a secondary outcome measure. Score range is 0-53, where low scores indicate low symptoms.
Changes in depressive symptoms (Beck) | 1 week, 2 weeks, 1 month
  Symptoms of depression will be measured before and after 5 sessions of tDCS using Beck Depression Inventory (BDI). Change BDI score will be used as a secondary outcome measure. Score range is 0-62, where low scores indicate low symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- CTI Northwestern, Chicago, Illinois, United States